CLINICAL TRIAL: NCT00257855
Title: A Randomised Controlled Trial of Neuroprotection With Lamotrigine in Secondary Progressive Multiple Sclerosis: Single Centre, Phase 2 Trial
Brief Title: A Randomised Controlled Trial of Neuroprotection With Lamotrigine in Secondary Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-001949-42
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2009-02

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: Secondary Progressive Multiple Sclerosis; Neuroprotection; Axonal loss; Brain atrophy; MRI; Lamotrigine; Sodium Channel Blockers
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lamotrigine

SUMMARY:
A present there is no safe treatment for reducing rate at which disability worsens in people with secondary progressive multiple sclerosis. Recent research has suggested the possibility that drugs that act by blocking the entry of sodium into nerve cells can protect nerve fibres in the brain and spinal cord. In this trial, the investigators will test whether one such drug, called lamotrigine, can prevent damage to nerve fibres and reduce the rate at which MS worsens. The period of treatment in the trial will run for 2 years.

DETAILED DESCRIPTION:
At present, there is no safe, widely applicable treatment that is capable of reducing the rate at which disability advances in secondary progressive multiple sclerosis (SPMS). There is good evidence that the primary cause of disability is axonal degeneration within the CNS, so there is considerable interest in developing treatments which can protect axons from degeneration. Experimental work by members of our group has established that axons may degenerate upon exposure to the inflammatory mediator nitric oxide. The mechanism of the damage implies that protection might be afforded by the novel approach of partially blocking sodium channels, and our group and others have recently demonstrated that drugs including flecainide, phenytoin and lamotrigine can reduce axonal degeneration when optic nerves or spinal roots are exposed to nitric oxide, and in experimental autoimmune encephalomyelitis.

Aims: To assess whether the sodium channel blocker lamotrigine has a neuroprotective, disease modifying effect on a) the rate of axonal degeneration and b) the accumulation of disability in patients with SPMS.

Methodology: We propose to recruit 120 people with SPMS in whom progression rather than relapse is the major cause of increasing disability into a double blind parallel group controlled trial lasting two years in which random allocation would be made to receive treatment with either lamotrigine or placebo. We anticipate that patient recruitment, follow-up and trial management could be achieved readily across four proposed sites in London. The primary endpoint would be an effect of treatment on cerebral atrophy, which correlates with other MR markers of axonal loss, and which can be measured reliably and sensitively using recently developed MR techniques. The trial is powered to detect a 60% beneficial effect on the rate of development of cerebral atrophy. Secondary endpoints would include effects of treatment on spinal cord atrophy and on clinical measurements of impairment/disability. MR measures of brain volume and cervical spinal cord cross-sectional area and scores of clinical impairment/disability would be determined at entry, and then after 12 and 24 months. Brain volume would be measured additionally at 6 and 18 months. Clinical follow-up would occur every 3 months, and interim analysis is planned at 12 months.

Utilization of results: A phase 2 trial of sodium channel blockade in SPMS is timely, given recent advances arising from experimental and imaging work. A successful outcome would enable sufficiently powered phase 3 trials to be implemented, but perhaps more significantly would demonstrate a novel, safe neuroprotective strategy to reduce long-term disability in this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60
* Progression rather than clinical relapse is the major cause for increased disability over the preceding 2 years
* EDSS 4.0-6.5

Exclusion Criteria:

* Very rapid deterioration in EDSS, >2 points over 6 months
* Use of Mitoxantrone in the preceding year
* Use of sodium channel blockers or calcium channel blockers in the preceding 2 weeks
* Use of corticosteroids in preceding 2 months
* Use of neuroprotective agents or immunosuppressants in the preceding 6 months
* Evidence of significant hepatic or renal impairment either in clinical history or blood results.
* Prior untoward reactions to lamotrigine, or severe temperature dependent symptoms
* Contraindications to MRI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Start 2005-11; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change in central brain volume on MRI using the 'Loseff method'

SECONDARY OUTCOMES:
Change in whole brain volume on MRI using Brain Boundary Shift Integral
Number and volume of new T2 high intensity lesion volume on T2 weighted MRI
Number and volume of new T1 low signal lesion volume on T1 weighted MRI
Ratio of new T1 to new T2 lesions on MRI
Change in magnetisation transfer ratio in normal MRI normal appearing white matter and normal appearing grey matter.
Change in upper cervical cord cross sectional area using the 'Loseff method' on MRI
Change in Kurtzke's Extended Disability Scaling Score.
Change in Multiple Sclerosis Functional Composite.
Change in Multiple Sclerosis Impact Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Raju Kapoor, MD PhD, Study Director — National Hospital for Neurology and Neurosurgery
Locations (1):
- National Hospital for Neurology and Neurosurgery, London, United Kingdom

REFERENCES:
- [Derived] Kapoor R, Furby J, Hayton T, Smith KJ, Altmann DR, Brenner R, Chataway J, Hughes RA, Miller DH. Lamotrigine for neuroprotection in secondary progressive multiple sclerosis: a randomised, double-blind, placebo-controlled, parallel-group trial. Lancet Neurol. 2010 Jul;9(7):681-8. doi: 10.1016/S1474-4422(10)70131-9. Epub 2010 Jun 8. PMID 20621711